CLINICAL TRIAL: NCT06720662
Title: Effect of Icosapent-ethyl Ester (IPE) to Reduce the Residual Risk in Patients Undergoing Secondary Prevention for Cardiovascular Disease.
Brief Title: Effect of Icosapent-ethyl Ester (IPE) to Reduce the Residual Risk Cardiovascular Disease.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Inar Castro Erger, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 77740424.3.3001.0068
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Atherosclerosis Cardiovascular Disease
Keywords: omega 3 fatty acids; atherosclerosis; oxylipins
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPE Supplementation Group (Active Comparator): Dietary Supplement: Icosapent Ethy capsules
  Interventions: Dietary Supplement: Icosapent-ethyl ester capsules
- Placebo Group (Placebo Comparator): Dietary Supplement: Corn oil Control
  Interventions: Dietary Supplement: Corn oil Control

INTERVENTIONS:
Dietary Supplement: Icosapent-ethyl ester capsules — Icosapent-ethyl ester (4.0 g of EPA) taken twice a day (2.0 g/day x 2) for six months.
  Arms: IPE Supplementation Group
Dietary Supplement: Corn oil Control — Corn oil twice a day (2.0 g/day x 2) for six months.
  Arms: Placebo Group

SUMMARY:
Cardiovascular diseases (CVDs) are the leading cause of global mortality, despite significant advances in prevention and treatment. Atherosclerosis, a chronic inflammatory condition, underlies ischemic events such as infarction and stroke, triggered by the instability and rupture of plaques. Current guidelines recommend drugs primarily aimed at reducing Low-Density-Lipoprotein cholesterol (LDL-C), arterial pressure, and glucose levels for atherosclerosis patients. However, there is little option of approved medications specifically targeting inflammation within the arterial plaques. Consequently, a significant proportion of patients face residual risks. On the contrary, numerous studies have highlighted the anti-inflammatory effects provided by omega-3 fatty acids (n-3 FA), specially the eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), and their derived oxylipins. These molecules exhibit the ability to enhance the phenotype of macrophages, increasing their capacity for efferocytosis, thereby improving plaque stability. Icosapent ethyl (IPE) is an esterifed version of eicosapentaenoic acid (EPA) and acts as a prodrug in the body to exert its effects. Icosapent ethyl (IPE) was the first fish oil product approved by the US Food and Drug Administration (FDA) to reduce the risk of atherosclerotic cardiovascular disease (ASCVD) in adults. Hence, the hypothesis of this study is that supplementing patients with IPE, in addition to their standard clinical treatment, will enhance macrophage functionality, thereby reducing inflammatory and oxidative stress biomarkers in comparison to a placebo. To test this hypothesis,a Randomized, Double-blind, Placebo-controlled Clinical trial will be performed, in which 294 patients under secondary prevention for CVDs will receive a 6-month supplementation of purified eicosapentaenoic acid-icosapent ethyl (4.0 g) daily or a Placebo (corn oil). Blood samples and anthropometric measurements will be taken at the beginning and end of the period. Basic clinical markers will be assessed, and monocytes will be collected and characterized. Fatty acid profiles and oxylipins will be determined through chromatography coupled with mass spectrometry. Finally, changes in biomarkers for both groups will undergo multivariate analysis to identify characteristics associated with the response to supplementation. Data from this study aims to provide support for physicians considering the prescription of bioactive compounds as a complementary therapy for atherosclerosis, with the goal of reducing residual risks and subsequently decreasing mortality resulting from cardiovascular events.

DETAILED DESCRIPTION:
A Randomized, Double-blind, Parallel, Placebo-controlled Clinical trial will be carried out. Initially, subjects will be randomly assigned to receive the supplementation or placebo treatment for 6 months. Daily supplemental treatment (IPE) will consist of Icosapent Ethy capsules (4.0 g of EPA) taken twice a day (2.0 g/day x 2). Placebo treatment (PLACEBO) will consist of similar capsules containing corn oil instead of IPE. It has been argued that the CV benefit with IPE in certain trials (most notably REDUCEIT) related to the use of pharmaceutical grade mineral oil as comparator (Sherratt et al., 2023). Although a comprehensive review of mineral oil use in CV trials found no reproducible, consistently statistically significant effect of mineral oil on inflammatory markers, including hsCRP (Olshansky et al., 2020), the investigators opted for use of corn oil as placebo, while there is no consensus about this subject. Participants will be instructed to consume half capsules after lunch and half after dinner. During the trial, the subjects will maintain their habitual routine and diet. Prescribed drugs will be kept without any change throughout the study. The Icosapent-ethyl (IPE) will be purchased from BASF S.A., Avenida Nacoes Unidas, 14171, 04794-000 Sao Paulo, Brazil, and the oil will be encapsulated in a Brazilian company still not defined.

ELIGIBILITY:
Inclusion Criteria: individuals from both sexes, aging 45 years or older having established CVD, without contraindications to the use of IPE, receiving a stable dose of a statin (± ezetimibe) for ≥4 weeks. Women should be not pregnant, not breastfeeding, not planning on becoming pregnant, and using an acceptable form of birth control during the study (if of child-bearing potential). Biomarkers should be:

hsCRP level - mg/liter: from 1 to 4.5; Triglyceride level - mg/dl: from 150 - 500; HDL cholesterol level - mg/dl: from 30 - 50 and LDL cholesterol level - mg/dl: from 40 - 100.

Exclusion Criteria: Patients with severe heart failure, active severe liver disease, a glycated hemoglobin level greater than 10.0%, a planned coronary intervention or surgery, a history of acute or chronic pancreatitis, or known hypersensitivity to fish, shellfish, or ingredients of icosapent ethyl or placebo. Autoimmune disease requiring the use of immunosuppressive therapy or current use of systemic corticosteroid therapy; Active neoplasm with indication for surgery, chemotherapy or radiation in the last 12 months (patients with a history of neoplasia and who have undergone curative surgery without the need for treatment in the last 12 months will be allowed); Inflammatory bowel disease or chronic diarrhea; Clinically significant non-transient hematological abnormalities; Renal dysfunction (GFR < 30 mL/min/1.73 m² and/or serum creatinine > 2.5 mg/dL or < 220 μmol/l); Severe liver disease (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] > 3x ULN in the last 6 months); Inability to sign the free and informed consent form; Participation in another clinical trial involving an investigational agent within 90 days prior to screening; Intolerance or hypersensitivity to statin therapy; History of acute or chronic pancreatitis; Malabsorption syndrome and/or chronic diarrhea; Use of non-study drug-related, non-statin, lipid-altering medications, dietary supplements, Niacin (>200 mg/d) or fibrates (unless ≥28-day washout). Any n-3 fatty acid medications (unless ≥28-day washout). Bile acid sequestrants (unless ≥7-day washout), PCSK9 inhibitors (unless ≥90-day washout); Other medications (not indicated for lipid alteration): Tamoxifen, estrogens, progestins, thyroid hormone therapy, systemic corticosteroids (local, topical, inhalation, or nasal corticosteroids are allowed), HIV-protease inhibitors that have not been stable for ≥28 days prior to the qualifying lipid measurements (TG and LDL-C) during screening. Cyclophosphamide or systemic retinoids during the screening period (unless ≥28- day washout) and/or plans for use during the treatment/follow-up period ; HIV-positive patients even without AIDS; Requirement for peritoneal dialysis or hemodialysis for renal insufficiency or creatinine clearance 5 × ULN or elevation due to known muscle disease; Drug or alcohol abuse within the past 6 months, and inability/unwillingness to abstain from drug abuse and excessive alcohol consumption during the study; 16 Mental/psychological impairment or any other reason to expect patient difficulty in complying with the requirements of the study or understanding the goal and potential risks of participating in the study.

Patients with Atrial fibrillation and Bleeding related disorders.

-

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Eicosapent ethyl ester (IPE) and high sensitivity C-Reactive Protein (hs-CRP) | From enrollment to the end of treatment at 6 weeks
  Eicosapent ethyl ester (IPE) combined with a classical pharmacological treatment, will contribute to reduce high sensitivity C-Reactive Protein (hs-CRP) in patients undergoing secondary prevention for cardiovascular disease.
  the concentration hsCRP was chosen based on the fact that it is the only inflammatory marker mentioned in the Prevention Guidelines (Arnett et al., 2019), was selected in the "Cantos" study (Ridker et al., 2018), has shown correlation with IPE in the "REDUCE-IT" study (Bhatt et al., 2019) and also having observed a reduction in patients supplemented with fish oil in other studies (Scolaro et al., 2018; Elisia et al., 2022).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cartolano FC, Dias GD, Miyamoto S, Damasceno NRT. Omega-3 Fatty Acids Improve Functionality of High-Density Lipoprotein in Individuals With High Cardiovascular Risk: A Randomized, Parallel, Controlled and Double-Blind Clinical Trial. Front Nutr. 2022 Feb 23;8:767535. doi: 10.3389/fnut.2021.767535. eCollection 2021. PMID 35281761
- [Background] Atar D, Jukema JW, Molemans B, Taub PR, Goto S, Mach F, CerezoOlmos C, Underberg J, Keech A, Tokgozoglu L, Bonaca MP. New cardiovascular prevention guidelines: How to optimally manage dyslipidaemia and cardiovascular risk in 2021 in patients needing secondary prevention? Atherosclerosis. 2021 Feb;319:51-61. doi: 10.1016/j.atherosclerosis.2020.12.013. Epub 2021 Jan 18. PMID 33476944
- [Background] Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Ballantyne CM; REDUCE-IT Investigators. Cardiovascular Risk Reduction with Icosapent Ethyl for Hypertriglyceridemia. N Engl J Med. 2019 Jan 3;380(1):11-22. doi: 10.1056/NEJMoa1812792. Epub 2018 Nov 10. PMID 30415628